CLINICAL TRIAL: NCT04801264
Title: Diagnosis of Adenoid Cystic Carcinoma on 68Ga-PSMA-617 PET-CT and Therapy With 177Lu-EB-PSMA-617
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCHPSMAACC
Record Dates: First submitted 2021-02-23; First posted 2021-03-16 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Adenoid Cystic Carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — gallium 68 PSMA-11; 177Lu-EB-PSMA-617

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA, PET/CT and 177Lu-EB-PSMA-617 therapy (Experimental): All patients diagnosed with ACC underwent 68Ga-PSMA PET/CT scan. If the PET/CT showed high PSMA expression in tumor lesions of some patients, they would intravenously injected with the dose about 1.85GBq (50 mCi) of 177Lu-EB-PSMA-617 for therapy.
  Interventions: Drug: 68Ga-PSMA; Drug: 1.85GBq (50 mCi) of 177Lu-EB-PSMA-617

INTERVENTIONS:
Drug: 68Ga-PSMA — Intravenous injection of one dosage of 74-148 MBq (2-4 mCi) 68Ga-PSMA. Tracer doses of 68Ga-PSMA will be used to image lesions of adenoid cystic carcinoma by PET/CT.
  Other Names: 68Ga-prostate specific membrane antigen
Drug: 1.85GBq (50 mCi) of 177Lu-EB-PSMA-617 — Patients were intravenous injected with the dose about 1.85GBq (50 mCi) of 177Lu-EB-PSMA-617 every 8 weeks (±1 week) for a maximum of 3 cycles.

SUMMARY:
Adenoid cystic carcinoma (ACC) accounts for 24% of salivary gland malignant tumors, is characterized by frequent local recurrences and distant metastasis, mainly to lungs. Considering its origination from salivary glands, an organ with intense physiological uptake of 68Ga-PSMA-617, this study aims to evaluate 68Ga-PSMA-617 uptake in local recurrent or metastatic ACC in comparison with 18F-FDG uptake in the same patients, and assess the feasibility of 177Lu-EB-PSMA-617 treatment in patients with the advanced ACC.

DETAILED DESCRIPTION:
Adenoid cystic carcinoma (ACC) is a rare tumor entity with a yearly incidence of 3-5 cases per million. ACC arises in the major salivary glands and more often in the minor salivary glands of the oropharynx, lip, nasopharynx, oral cavity, nasal cavity, paranasal sinus, larynx and tracheobronchial tree. ACC is characterized by frequent local recurrences and distant metastasis, mainly to lungs. 18F-FDG PET/CT is considered to be a viable tool to assess ACC at initial presentation. However, FDG uptake in ACC is lower than in squamous cell carcinoma (SCC) and not all ACC lesions show detectable FDG uptake. So, it is necessary to find another effective way to detect ACC and its metastases. As in known, PSMA is highly expressed in salivary glands, and Wim van Boxtel et al had demonstrated high PSMA-ligand uptake in a patient with recurrent and metastatic ACC using 68Ga-PSMA PET/CT. 68Ga-PSMA has been developed as a targeting imaging agent widely used in prostate cancer in prostate cancer. Thus, this prospective study is going to investigate whether 68Ga-PSMA PET/CT may be superior for diagnosis, therapy response assessment and follow-up of ACC than 18F-FDG PET/CT. Furthermore, peptide receptor radionuclide therapy has been widely used in the treatment of prostate cancer lesions that showed high PSMA uptake on 68Ga-PSMA PET/CT, we'll try to assess the safety and therapeutic response to 177Lu-EB-PSMA-617 in patients with ACC.

ELIGIBILITY:
Inclusion Criteria:

* confirmed treated or untreated adenoid cystic carcinoma patients;
* 18F-FDG PET/CT within two weeks;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* known allergy against PSMA
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 1 year
  Sensitivity and Specificity of 68Ga-PSMA PET/CT for adenoid cystic carcinoma in comparison with 18F-FDG PET/CT

SECONDARY OUTCOMES:
Safety of therapy | through study completion, an average of 1 year
  the safety assessed by CTCAE v4.0

OTHER OUTCOMES:
Therapeutic effect | through study completion, an average of 1 year
  the therapeutic response assessed by PSMA PET/CT to 177Lu-EB-PSMA-617 in patients with adenoid cystic carcinoma.
Correlation between PSMA expression and SUV in PET/CT | through study completion, an average of 1 year
  to mearsure the SUVmax of ACC on PSMA PET/CT and to investigate the expression of PSMA on primary, recurrent and metastatic ACC tumour tissue using immunohistochemistry, and analyze the correlation between them.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang G, Zhou M, Zang J, Jiang Y, Chen X, Zhu Z, Chen X. A pilot study of 68 Ga-PSMA-617 PET/CT imaging and 177Lu-EB-PSMA-617 radioligand therapy in patients with adenoid cystic carcinoma. EJNMMI Res. 2022 Aug 19;12(1):52. doi: 10.1186/s13550-022-00922-x. PMID 35984529